CLINICAL TRIAL: NCT06535035
Title: Evaluation of the Analgesic and Anti-Inflammatory Impact of Photobiomodulation in Patients With Dental Implants
Acronym: AAPDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Professor Oral Medicine, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2934/2020
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Dental Pain and Sensation Disorder
Keywords: laser; pain, dental implant , quality of life , MDA
MeSH Terms: conditions — Toothache; Sensation Disorders; Pain | interventions — Laser Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: During the initial evaluation, data collection, informed consent, a complete clinical and oral evaluation, as well as a radiological study with cone beam computed tomography (CBCT) were carried out. Subsequently, surgical intervention was performed with the placement of dental implants. In the experimental group, low-level laser therapy (LLLT) was applied, while a placebo procedure (SHAM) was used in the control group. Pain and inflammation were evaluated using visual analog scales (VAS) from day 0 to 7 days postoperatively. Additionally, MDA levels were measured and the OHIP-14 questionnaire was used to assess oral health-related quality of life
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 laser therapy (Experimental): Data collection, informed consent, a complete clinical and oral evaluation, as well as a radiological study with cone beam computed tomography (CBCT). A surgical intervention was performed with the placement of dental implants. In the experimental group, low-level laser therapy (LLLT) was applied immediately after the placement of the implants in a single session with an EPIC X Biolase diode laser (BIOLASE, Inc., USA), voltage 100-240 V, 1.5 A, power 0.5 W, 10-20 J, for 10-30 seconds. It was applied to three points in the area: buccal side, palatal/lingual side, and occlusal side to stimulate the tissue.Pain and inflammation were evaluated using visual analog scales (VAS) from day 0 to 7 days postoperatively. Additionally, MDA levels were measured and the OHIP-14 questionnaire was used to assess oral health-related quality of life
  Interventions: Device: laser therapy After implant surgery, laser therapy (LLLT) was applied
- group Sham (Sham Comparator): data collection, informed consent, a complete clinical and oral evaluation, as well as a radiological study with cone beam computed tomography (CBCT). Surgical intervention was performed with the placement of dental implants. In the group sham comparate p, low-level laser therapy (LLLT) was applied inactive . Pain and inflammation were evaluated using visual analog scales (VAS) from day 0 to 7 days postoperatively. Additionally, MDA levels were measured and the OHIP-14 questionnaire was used to assess oral health-related quality of life
  Interventions: Device: SHAM

INTERVENTIONS:
Device: laser therapy After implant surgery, laser therapy (LLLT) was applied — After implant surgery, laser therapy (LLLT) was applied a single session with an EPIC X Biolase diode laser (BIOLASE, Inc., USA)
  Other Names: Experimental
  Arms: Group1 laser therapy
Device: SHAM — After implant surgery, After implant surgery, laser therapy (LLLT) was applied in the same manner but without activating it
  Other Names: After implant surgery, laser therapy (LLLT) was applied without activating it
  Arms: group Sham

SUMMARY:
The aim of this study is to evaluate the analgesic and anti-inflammatory effects of photobiomodulation in participants undergoing dental implant placement.

A randomized clinical trial was conducted with 62 participants requiring dental implant placement, divided into two groups of 31 each. Immediately after implant placement, one group received diode laser photobiomodulation, while the SHAM group received sham treatment. Pain and inflammation were assessed at 24 h, 48 h, and 7 days. In addition, Modified Dental Anxiety (MDA) levels were measured and the Oral Health Impact Profile-14 (OHIP-14) questionnaire was used to assess oral health-related quality of life.

DETAILED DESCRIPTION:
Low-Level Laser Therapy (LLLT) has revolutionized medicine, promoting the healing and regeneration of tissues in an innovative way. This study focuses on evaluating the powerful analgesic and anti-inflammatory effects of LLLT in patients undergoing dental implant placement.

Methodology A randomized clinical trial was conducted with 62 patients, divided into two groups of 31 each. One group received photobiomodulation with a combined 630 and 808 nm diode laser, while the SHAM group received a simulated treatment.

Inclusion criteria: Participants who needed dental implant rehabilitation and signed the informed consent. Participants with a poor general health status, decompensated chronic diseases (diabetes) , pregnant women, and those with bleeding disorders were excluded.

Procedure:

Informed consent, data collection, complete clinical and oral evaluation, and radiological study with CBCT.

Surgical intervention:

Placement of dental implants. In the experimental group, low-level laser therapy (LLLT) was applied immediately after the placement of the implants in a single session with an EPIC X Biolase diode laser (BIOLASE, Inc., USA), voltage 100-240 V, 1.5 A, power 0.5 W, 10-20 J, for 10-30 seconds. It was applied to three points in the area: buccal side, palatal/lingual side, and occlusal side to stimulate the tissue.

Pain and inflammation were evaluated using visual analog scales (VAS) from day 0 to 7 days postoperatively. Additionally, MDA levels were measured and the OHIP-14 questionnaire was used to assess oral health-related quality of life

ELIGIBILITY:
Inclusion Criteria:

* Participants who needed dental implant rehabilitation and signed the informed consent

Exclusion Criteria:

* Participants with a poor general health status, decompensated chronic diseases, pregnant women, and those with bleeding disorders were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Pain levels assessed with the visual analogue scale (VAS) | 24h-48h,7 days
  A score of 0 indicated no pain while 10 indicated the worst pain possible
inflammation evels assessed with the visual analogue scale | 24h-48h,7 days
  A score of 0 indicated no inflammation while 10 indicated the worst inflammation possible

SECONDARY OUTCOMES:
Modified Corah Dental Anxiety Scale (MDAS) | at day 0 and 7 days
  (0 relaxed, 1 slightly anxious, 2 quite anxious, 3 very anxious or 4 extremely anxious). The total sum was obtained and 4 ranges of fear and anxiety were established (<9 mild or no anxiety, 9-12 moderate anxiety, 13-14 high anxiety, >14 phobic anxiety, >14 very anxious anxiety, >14 very anxious anxiety, >14 very anxious anxiety, >14 very anxious anxiety, >14 very anxious anxiety).
OHIP-14sp | at 0 and at 7 days
  consists of 14 questions related to different dimensions of the patient's quality of life (functional limitation, pain, psychological problems, etc.) higher score worse quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

REFERENCES:
- [Background] Qu C, Luo F, Hong G, Wan Q. Effects of photobiomodulation therapy on implant stability and postoperative recovery: a systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2022 Jun;60(5):e712-e721. doi: 10.1016/j.bjoms.2022.01.014. Epub 2022 Feb 5. PMID 35490059
- [Background] Heidari M, Paknejad M, Jamali R, Nokhbatolfoghahaei H, Fekrazad R, Moslemi N. Effect of laser photobiomodulation on wound healing and postoperative pain following free gingival graft: A split-mouth triple-blind randomized controlled clinical trial. J Photochem Photobiol B. 2017 Jul;172:109-114. doi: 10.1016/j.jphotobiol.2017.05.022. Epub 2017 May 18. PMID 28549319